CLINICAL TRIAL: NCT03359109
Title: Effect of Metallosis on Tissues and Serum Metal Levels in Children With Orthopedic Implants
Brief Title: Metallosis on Tissues and Serum Metal Levels in Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, A. Noelle Larson, MD, Associate Professor of Orthopedics, Mayo Clinic
Other Study IDs: 17-004970
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Orthopedic Disorder; Retained Metal Implant
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Waste Surgical Tissue, possible cell-line development

GROUPS / COHORTS (3):
- Stainless Steel Devices: 10 patients with stainless steel devices implanted
- Titanium or Titanium-alloy Based Devices: 30 patients with titanium or titanium-alloy implanted devices
- De Novo Titanium Implant: 10 patients undergoing de novo titanium implant placement who have had no previous orthopedic procedures

SUMMARY:
Slightly elevated blood metal levels have been found in adults undergoing hip and knee replacement. It is unknown whether pediatric patients with metal implant(plates/screws/rods) have elevated blood metal levels. This may have an impact on practice if children have high blood metal levels with routine orthopedic implants. If researchers find elevated metal levels, they may recommend patients to have the plates removed or may switch to a different type of metal. Further work on this topic is needed.

DETAILED DESCRIPTION:
Metal implants are routinely placed in children for treatment of fracture or deformity. Long-term effects of indwelling metal implants are not well-understood. Data from this study will provide guidances as to whether some metals are safer for children (stainless vs. titanium alloys). In addition, we will document the presence of serum ion concentration for children with metal implants in place and whether this resolves after implant removal. Tissues adjacent to implants will be evaluated for signs of metallosis and wear debris. Presence of metallosis will be correlated with serum ion concentration. In vivo studies will provide data on whether metal exposure to bone cells and fibroblasts affects their inflammatory cascade and function. Based on these findings, surgeons can better counsel patients whether routine implant removal is advisable or whether stainless steel implants are safer for long-term retention compared to titanium implants. Further, novel drug targets for treatment and prevention of metallosis will be developed. This project will foster collaboration and future partnerships between the Sanford Health and Mayo Clinic research teams

ELIGIBILITY:
Inclusion Criteria:

* Ages 4 years - 18 years
* Stainless steel, titanium or titanium-alloy based implants, scheduled for surgery
* De novo surgery where titanium implant placement

Exclusion Criteria:

* Concomitant infection

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing orthopedic surgery to remove or place metal implants.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mechanistic responses of bone repair cells upon Ti exposure | 3-6 months
  To address how deregulated bone repair provokes adverse reactions, the investigators will monitor gene regulatory effects in cell culture models of titanium exposure by either silencing or activating key biological pathways

SECONDARY OUTCOMES:
Evaluate serum levels of metal ions | 3-6 months
  To evaluate systemic effects of metal ions on children, the investigators will determine whether metal ion levels are elevated in participants with retained implants by intraoperatively blood draw and at first postoperatively visit. Conversely, participants undergoing implant placement will also have ion levels taken intraoperatively and then at latest follow-up visit to see if implants cause in increase in serum metal levels

CONTACTS AND LOCATIONS:
Overall Officials: A.Noelle Larson, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials